CLINICAL TRIAL: NCT01574586
Title: A Multicenter, Randomized Trial to Compare 2 Link Nobori and 3 Link Xience Stents in Bifurcation Stenting
Brief Title: Bifurcation Stenting Using 2 Link Stent Nobori Versus 3 Link Stent Xience
Acronym: BEGIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Kurashiki Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BEGIN12
Record Dates: First submitted 2012-04-06; First posted 2012-04-10 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Stenosis
Keywords: True Bifurcation stenosis
MeSH Terms: conditions — Coronary Stenosis

ARMS (2):
- 2-link stent Nobori (Active Comparator): Bifurcation stenting
  Interventions: Device: Bifurcation stenting
- 3-link stent Xience (Active Comparator): Bifurcation stenting
  Interventions: Device: Bifurcation stenting

INTERVENTIONS:
Device: Bifurcation stenting — Bifurcation stenting using 2-link stent Nobori versus 3-link stent Xience

SUMMARY:
The primary objective of this study is to make a comparison of safety and efficacy of DESs with different link number (2-link Nobori and 3-link Xience) in patients with de novo true bifurcation lesions.

The minimum lumen diameter of the side branch ostium in bifurcation at 8 months and the MACE rate until one year after PCI will be assessed in both groups.

ELIGIBILITY:
Inclusion Criteria:

1. Patient eligible for percutaneous coronary intervention
2. Patient or substitute decision-maker willing to provide written informed consent, which is approved by the Institutional Review Board or its equivalence
3. De novo stenosis at coronary bifurcation with up to two vessels (visually estimated diameter stenosis ≥50%)
4. Second vessel at coronary bifurcation treatable with trial device during the procedure
5. True coronary bifurcation, ≥50% diameter stenosis in both the main and side branches, belonging to the Medina classes 1.1.1, 1.0.1, and 0.1.1,
6. Visually estimated target lesion reference vessel diameter, 2.5-5.0 mm in the main branch, ≥2.25 mm in the side branch
7. Target lesion treatable with one or two stents in both the main and side branches
8. Consensus of PCI after discussion between cardiologists and cardiac surgeons for the lesion in the left main coronary artery
9. Thrombolysis in Myocardial Infarction grade ≥1 flow in both the main and side branches

Exclusion Criteria:

A. General restrictions

1. Unable to be followed by the implementing medial institution
2. Life expectancy <1 year
3. Acute myocardial infarction (<1 week)
4. Left ventricular ejection fraction <30%
5. Scheduled for elective treatment requiring antiplatelet drug Withdrawal
6. Deemed as unsuitable by the investigator or subinvestigator
7. Serum creatinine level ≥2.0 Mg/dl

B. Vascular morphological restrictions

1. Lesion proximal to coronary artery bypass graft anastomotic site (visual estimation ≤5.0 mm) or including a part of coronary artery bypass grafting
2. In-stent restenosis
3. Severe calcification

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-05 (Actual); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
Minimum lumen diameter of the side branch ostium in bifurcation | 8 months

SECONDARY OUTCOMES:
Incidence of MACE | in-hospital, 30 days, 8 months, 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Kurashiki Central Hospital, Kurashiki, Japan